CLINICAL TRIAL: NCT06883708
Title: iSupport-Malaysia: An Online Psychoeducational Intervention Program for Informal Dementia Caregivers in Malaysia - A Pilot Feasibility Study
Brief Title: Feasibility & Preliminary Impacts of an Online Psychoeducational Program (iSupport-Malaysia) for Informal Dementia Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunway University (Other)
Collaborators: Sarawak General Hospital (Other); Sarawak Heart Centre (Other); University of Malaya (Other)
Responsible Party: Principal Investigator, Ken Joey Loh, Clinical Psychologist & PhD Candidate, Sunway University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: iSupport-Malaysia 2024/REC0133; NMRR-ID-24-01472-ZAI (Other: Medical Research & Ethics Committee, Ministry of Health Malaysia); MRECID 202499-14190 (Other: Medical Research Ethics Committee, Universiti Malaya Medical Center, Malaysia)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Caregiver Subjective Burden; Caregiver Wellbeing; Feasibility Pilot Study
Keywords: informal caregivers; dementia; caregiver support; internet-based intervention; psychoeducation
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Experimental parallel between-group design with two arms
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants are aware of the intervention they receive (web program or eBook).
  Nonetheless, site investigators involved in recruitment are blinded to the randomisation sequence. The data analyst will also be blinded to the intervention assigned to the participants, as all participants' data are labelled using universal subject IDs that do not distinguish between groups of participants. Data collection of baseline and post-intervention assessments will be self-administered online by the participants and remain anonymous. Hence, researchers have no influence over the outcomes of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- iSupport-Malaysia Web-Based Intervention (Experimental): Access to the online, web-based version of iSupport-Malaysia throughout the 3-month study period. The 23 lessons will be arranged under the 5 modules in the same way as the original iSupport manual. Each lesson will be delivered in bite-sized knowledge, using engaging videos, interactive quizzes with feedback, and reflection exercises. Each lesson will take an average of 10-20 minutes to complete. At the end of each lesson, a completion batch will be given. The lesson plan can be personalised by the caregivers themselves according to individual needs. Caregivers will also have the option to receive a course completion certificate if they successfully completed all 23 lessons in the program.
  Additionally, in each lesson, participants are encouraged to post comments in response to the prompt questions, and also reply to others' comments.
  Interventions: Behavioral: iSupport-Malaysia Web-Based Intervention
- iSupport-Malaysia eBook (Active Comparator): Receive the Malay-translated, culturally adapted version of the 'iSupport for Dementia' manual in PDF format throughout the 3-month study period. This eBook is approximately 275 pages long, containing comprehensive text-based details for the 5 modules and 23 lessons. The modules and lessons are similar to the iSupport-Malaysia web-based program. Each lesson includes at least one case 1 scenario(s) presented in a quiz format. Some lessons offer additional worksheets for caregivers to reflect on their own caregiving experiences and apply the strategies learned to their caregiving journey. A completion batch is given at the end of each lesson. The lesson plan can be personalised by the caregivers themselves according to individual needs.
  Interventions: Behavioral: iSupport-Malaysia eBook

INTERVENTIONS:
Behavioral: iSupport-Malaysia Web-Based Intervention — iSupport-Malaysia web-based intervention is a website version of the culturally adapted "iSupport for Dementia" into the Malaysia context (in local Malay language).
  The 23 lessons is arranged under the 5 modules in the same way as the original iSupport manual. Each lesson is delivered in bite-sized knowledge, using engaging videos, interactive quizzes with feedback, and reflection exercises. Each lesson takes an average of 10-20 minutes to complete. At the end of each lesson, a completion batch is given. The lesson plan can be personalised by the caregivers themselves according to individual needs. Caregivers will also have the option to receive a course completion certificate if they completed all 23 lessons in the program. Additionally, in each lesson, participants are encouraged to post comments in response to the prompt questions, and also reply to others' comments.
  Arms: iSupport-Malaysia Web-Based Intervention
Behavioral: iSupport-Malaysia eBook — iSupport-Malaysia eBook is the Malay-translated, culturally adapted version of the "iSupport for Dementia" manual in PDF format. This eBook is approximately 275 pages long, containing comprehensive text-based details for the 5 modules and 23 lessons. The modules and lessons are similar to the iSupport-Malaysia web-based program. The main lesson content is delivered in text-based format. Each lesson includes at least one case 1 scenario(s) presented in a quiz format. Some lessons offer additional worksheets for caregivers to reflect on their own caregiving experiences and apply the strategies learned to their caregiving journey. A completion batch is given at the end of each lesson. The lesson plan can be personalised by the caregivers themselves according to individual needs.
  Arms: iSupport-Malaysia eBook

SUMMARY:
The general objective of this pilot feasibility study is to implement the pilot randomised controlled trial (RCT) and evaluate the feasibility of its methods and procedures for iSupport-Malaysia intervention. Another objective is to assess the acceptability and preliminary impacts of the iSupport-Malaysia web-based intervention on the psychological well-being of informal caregivers (ICs) of persons living with dementia (PLWDs) in Malaysia, compared to iSupport-Malaysia eBook.

The main questions this pilot study aims to answer are:

1. How feasible is it to implement iSupport-Malaysia as an accessible resource for ICs of PLWD in Malaysia?
2. Does the use of iSupport-Malaysia lead to a reduction in caregiver burden among the ICs of PLWD in both web and eBook conditions?
3. Does the use of iSupport-Malaysia lead to improvements in psychological well-being (e.g. reduced depression, anxiety, stress; and increased quality of life) among the ICs of PLWD in both web and eBook conditions?
4. What are the perceptions of ICs of PLWD on the usability, satisfaction and perceived usefulness of the modules in iSupport-Malaysia?

To answer these research questions:

Seventy ICs of PLWD who met the study criteria will be recruited from the geriatric facilities of three hospitals, as well as via social media and referrals from elderly care centres.

Eligible participants will sign an informed consent form, and be randomly assigned to the intervention (iSupport-Malaysia web program) or active comparison group (iSupport-Malaysia eBook) using stratified block randomisation.

In both arms, participants are required to complete at least 10 out of 23 lessons within 3 months.

Outcome measures will be administered online at baseline, 1-month and 3-month follow-up.

Feasibility outcomes will also be measured. Upon completion of the program, ICs in the experimental group will be invited for in-depth interviews via an online teleconferencing platform.

Expected outputs:

A free, adaptive web-based iSupport-Malaysia in the local Malay language. iSupport-Malaysia can facilitate self-directed training in public and private dementia services, integrate into caregiver training programs, and promote self-directed public education on dementia care.

DETAILED DESCRIPTION:
BACKGROUND

Informal caregivers (ICs) refer to family members who provide unpaid physical and psychological care to their relatives affected by chronic illnesses, including dementia. Caregiving responsibilities often include assisting in activities of daily living (ADLs) of the PLWD, managing medication, as well as providing emotional support to the PLWDs. A recent systematic review revealed that Malaysian ICs of PLWD often experienced moderate to high burden in their caregiving roles due to not knowing how to manage the BPSDs; aside from limited psychosocial support, awareness and education (Mohd Razi et al., 2023).

While face-to-face dementia caregiver training programs have shown benefits, their implementation in low- and middle-income countries (LMICs) faces challenges due to limited awareness, funding, and infrastructure (Pot et al., 2019). Hence, internet-based caregiver interventions may offer a solution to reach more caregivers and increase service coverage. With internet users comprising 96.0% of the total population in Malaysia (98.1% in urban, 89.1% in rural; Department of Statistics, 2022), an online intervention is deemed suitable in the Malaysian context.

To the best of the authors' knowledge, only two interventional studies have been published locally for ICs of PLWD. Hence, the current iSupport study might be one of the first local research studies to evaluate the feasibility, acceptability and preliminary impacts of a digital intervention program on the psychological well-being of ICs of PLWD in Malaysia.

RELATED WORK (PHASE 1 STUDY)

The investigators have obtained permission from the WHO to culturally adapt "iSupport for Dementia"© into the local Malaysian context. Upon professional translation of all texts in the generic iSupport into the local Malay language, all content in the eBook has been adapted into short educational videos. These videos, interactive quizzes, and reflection exercises were then hosted on a Learning Management System (LMS) platform, creating the iSupport-Malaysia web-based intervention program.

The first two web prototypes were evaluated critically by conducting focus groups and usability testing sessions with stakeholders (healthcare professionals, formal and informal caregivers of PLWD). Feedback obtained from these sessions was used to improve the content and user interface of the web prototype. Content validation was also performed via quantitative and qualitative appraisals, as well as fidelity checks by the program authors from the WHO.

At the time of writing, the Phase 1 study data collection has been completed. The current study protocol focuses on the Phase 2 Pilot Feasibility Study.

METHODOLOGY

STUDY DESIGN:

This is an experimental pilot feasibility study adopting mixed-methods, two-arm parallel randomised controlled design.

Eligible ICs of PLWD will be randomised (1:1 ratio) into either: (1) iSupport-Malaysia web-based intervention; or (2) iSupport-Malaysia eBook.

Web intervention group will be given access to the iSupport-Malaysia website throughout the study period. The eBook comparison group will be provided with iSupport-Malaysia eBook throughout the study period. After the intervention ends, both groups will receive access to both the website and eBook.

Study duration per participant is 3 months. Assessments on psychological wellbeing are administered pre-measurement (t0), first follow-up (t1, 1 month after t0), and second follow-up (t2, 3 months after t0). Data will be collected online via secured REDCap platform.

RANDOMISATION:

Stratified block randomisation will be used to randomly assign eligible, consented participants to either the web intervention or eBook condition.

First, participants will be stratified by gender (male or female); and relationship of the IC to the PLWD (child or non-child).

Then, participants will be randomised with 1:1 allocation using a block size of 2.

To prevent researcher bias, the randomisation tables for each striatum will be prepared by an independent researcher not involved in participant recruitment. The same independent researcher will provide the group allocation of the participants upon obtaining the enrolment list.

SAMPLE:

Study population:

All informal caregivers (ICs) who are currently taking care of a person living with dementia (PLWD). The ICs of PLWD included in this study are all self-reported adult family caregivers for dementia persons from Universiti Malaya Medical Centre (UMMC), Sarawak General Hospital (SGH), Sarawak Heart Centre (SHC), caregivers' support groups (online/ offline), and elderly care centres around the nation.

Sampling method:

Convenient sampling will be used for in-person recruitment at geriatric facilities at hospital sites (UMMC, SGH and SHC).

Volunteer sampling will be used for online recruitment from caregivers' support groups (online social media/ offline), and elderly care centres around the nation.

Sample size:

For a two-armed pilot trial, several rules of thumb have provided an estimation of the total sample size to range between 20 and 70.

Whitehead et al. (2016) recommended a sample size of 25 per treatment arm to achieve a power of 90%, two-sided significance of 0.05, and a small standardised effect size (0.1 < σ < 0.3).

Conservatively considering a dropout rate of 40% in this pilot study, a total of 70 ICs of PLWD will be recruited (35 per treatment arm).

DATA COLLECTION:

1. Screening Procedure:

   Hospital Sites: Site investigators at respective hospital sites will approach ICs of PLWD at the clinic waiting area or geriatric wards to explain the iSupport study. Interested ICs will fill up the pen-and-paper screening questionnaires on the spot.

   Other Sites: Investigators will post and circulate the study advertisement in English and Bahasa Malaysia on social media (caregivers' support groups on Facebook and WhatsApp), and elderly care centres contacts. Interested ICs will scan the QR code on the study poster to register their interest. Then, the investigator will contact the ICs and send a secured REDCap link to the online screening questionnaire.

   The screening questionnaires include: i) Brief demographic questionnaire assessing the inclusion & exclusion criteria; ii) Ascertain Dementia 8-item (AD8), Malay version; iii) 1-item burden scale; iv) Hospital Anxiety & Depression Scale (HADS), Malay version.
2. Informed Consent Procedure:

   Hospital Sites: Eligible ICs will be given the physical information sheet to read and ask questions about the study. If they agree to participate, they will sign the hardcopy informed consent form.

   Other Sites: Eligible ICs will be sent (via email or WhatsApp) the PDF version of the information sheet to read and ask questions about the study. If they agree to participate, they will insert their digital signature and return the signed consent form to the investigator. Once the signed consent form is downloaded to the investigator's password-protected personal computer, the investigator will delete the consent form copy from the email and WhatsApp chat (to protect participants' privacy in the event of data breach).

   Consented participants will be told that they will receive their group allocation, secured questionnaire links and further instructions via email.

   Ineligible participants will not be invited to join the study. Nonetheless, the investigator will offer them the generic English version of the "iSupport for Dementia" eBook, and also an option of whether they would like to receive the culturally adapted version of iSupport eBook in Bahasa Malaysia after study closure. They will also be encouraged to speak to their healthcare providers and seek support from local dementia associations.
3. Baseline Measurement and Group Allocation:

   The enrolment list will be given to the independent researcher doing the randomisation, who shall then revert back to the P.I. about the group allocation of each consented participant.

   P.I. will email consented participants to inform them about their group allocation, and attach the secured link to complete the baseline questionnaires via REDCap.

   Participants can reach out to the investigator via phone, WhatsApp or email if they have any questions.
4. Procedure of Intervention:

   According to their group allocation, participants will receive access to either the iSupport-Malaysia website or the iSupport-Malaysia eBook throughout the study period.

   At 1 month and 3 months after randomisation, participants will be emailed secured links to complete the 1-month and 3-month follow-up assessments on REDCap.

   Finally, at the end of the 3-month intervention, selected participants from the web group will be invited to a virtual semi-structured interview (via Zoom) to gather their user experience and insights until data saturation is reached.
5. Treatment Compliance Protocol:

To ensure consistent 'dosage' and treatment effect, participants in both groups are encouraged to: i) use the iSupport at least once a week; ii) complete a minimum of 10 lessons at the end of the 3-month intervention program.

Email or WhatsApp reminders will be sent once per fortnight to encourage continuous usage.

Intervention adherence will be monitored during the 1-month and 3-month follow-up, where participants will be asked to self-report: i) whether they have used the iSupport every week for the past 1 month/ 3 months; ii) the average duration spent on iSupport every week; and iii) the total number of lessons completed in 1 month / 3 months respectively.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older, any gender
* Able to understand written Malay language
* A self-reported caregiver of person living with any form of dementia (defined by a score of ≥ 2 on the AD8)
* Provide unpaid care to the PLWD for at least 6 months at the time of recruitment
* Experience some extent of psychological distress, such that they should experience some levels of subjective burden (defined by a score of ≥ 4 on the 1-item burden scale ranging from 1 to 10), OR some symptoms of depression OR anxiety (defined by a score of ≥ 8 on either the 'depression' or 'anxiety' subscales of HADS)
* Regular internet user, defined as using the internet at least twice a week.

Exclusion Criteria:

* Already participated in Phase 1 iSupport-Malaysia studies (focus groups, usability testing)
* Where another family member in the same household has participated/ currently participating in the iSupport study
* Have limited comprehension of written Malay language
* Do not have access to a device with an internet connection (e.g. mobile phone, tablet, laptop, desktop) more than twice a week
* Unable or unwilling to provide written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | Screening
  Percentage of ICs who meet the eligibility criteria among all the screened ICs of PLWD.
Randomisation Feasibility | Baseline
  Percentage of ICs who agree to randomisation among all eligible ICs.
Retention Rates | 3 months
  Percentage of participants retained until the end of the study in both arms.
Program Engagement Rate | 3 months
  Percentage of ICs who comply to the treatment protocol in both arms.

SECONDARY OUTCOMES:
Zarit Burden Interview (ZBI), Malay version | Baseline, 1 month, 3 months
  Caregiver subjective burden will be measured using Zarit Burden Interview (ZBI), Malaysia validated version (in Malay language).
  The ZBI is a 22-item self-report questionnaire that measures subjective burden in caregivers. Items are rated on a 5-point scale from 0 (never) to 4 (almost always). Total scores range from 0 to 88, with higher scores indicating greater subjective burden.
  The total scores are categorised into: 0-20 (little or no burden), 21-40 (mild to moderate burden), 41-60 (moderate to severe burden), and 61-88 (severe burden). Nonetheless, the validation study in Malaysia suggested a score of 22 as the suitable cut-off score for M-ZBI scale in the local population. At this cut-off, the M-ZBI demonstrated 70.8% sensitivity and 69.2% specificity for detecting burden among Malaysian caregivers (Shim et al., 2018).
  Changes in subjective burden will be assessed by M-ZBI total scores from baseline to 1-month and 3-month follow-ups.
Hospital Anxiety & Depression Scale (HADS), Malay version | Baseline, 1 month, 3 months
  The HADS measures symptoms of anxiety and depression through total scores obtained on its respective 7-item subscales, using a 4-point scale each (Snaith & Zigmond, 1986). Subscale scores range from 0-21, with higher scores indicating more severe anxiety or depression. The Malaysia-validated version in Malay language will be administered.
  Changes in symptoms of depression and anxiety will be assessed by the HADS-D and HADS-A subscale scores from baseline to 1-month and 3-month follow-ups.
Perceived Stress Scale (PSS-10), Malay version | Baseline, 1 month, 3 months
  The 10-item PSS aims at assessing the extent to which an individual appraises life events as stressful (Cohen et al., 1983). This questionnaire requires the participants to rate the degree to which their lives had been unpredictable, uncontrollable and overloading for the past month. The items were designed on a five-point Likert scale, from 0 (never) to 4 (very often). Item responses will be summed after reverse-scoring four items, yielding a total score for perceived stress. The Malaysia-validated version in Malay language will be administered.
  Changes in perceived stress will be assessed by PSS-10 total scores from baseline to 1-month and 3-month follow-ups.
WHO Quality of Life, Brief Version (WHOQOL-BREF), Malay version | Baseline, 1 month, 3 months
  The WHOQOL-BREF assesses quality of life (QoL) through scores on four domains: physical health, psychological, social relationships and environment (The WHOQOL Group, 1998). Participants will be required to answer two general questions on overall QoL and health satisfaction; as well as 24 specific questions assessing physical health (7 items), psychological health (6 items), social relationships (3 items), and environment (8 items). Their experiences over the past two weeks will be rated on 5-point scale. This 26-item instrument will produce transformed scores from 0-100, with higher scores representing better QoL. The Malaysia-validated version in Malay language will be administered.
  Changes in quality-of-life scores will be assessed by WHOQoL-BREF total scores from baseline to 1-month and 3-month follow-ups.

OTHER OUTCOMES:
System Usability Scale (SUS), Malay version | 3 months
  The System Usability Scale (SUS) (Brooke, 1996) will be used to evaluate the usability of iSupport-Malaysia web-based program. Each statement in the questionnaire will be rated on a 5-point Likert scale of 0 (strongly agree) to 4 (strongly disagree). Total scores range from 0 to 40, and will be multiplied by 2.5 to convert the scores to 0-100. Higher scores indicate better usability of a website. The Malaysia-validated version in Malay language will be administered.
  Here, the SUS will be administered to the web-based intervention group upon study completion. A total score of 68 and above would indicate above average usability score of our iSupport-Malaysia web version of the intervention.
Ascertain Dementia 8-item (AD8), Malay version | Screening
  Ascertain Dementia 8-item (AD8) (Galvin et al., 2005) is a brief informant-based questionnaire used to screen for cognitive impairment and dementia. It consists of 8 questions that are answered by a reliable informant, such as a family member or close friend of the patient being evaluated. The informant will rate changes in the patient's memory, problem-solving abilities, orientation, daily activities, and adaptive functioning compared to a few years ago. Each item is answered by selecting one of the three options: "Yes, A Change", "No, No Change", or "N/A, Don't Know". The final score is the sum of the number of items answering "Yes, A Change". Total score ranges from 0 to 8, with higher scores indicating greater cognitive impairment.
  The Malaysia-validated version in Malay language will be administered. At screening, the cut-off score of 2 and above indicates that the care recipient has cognitive difficulties.
Sociodemographic Data | Screening, baseline
  General information about the ICs will be obtained: age, gender, ethnicity, religion, occupation, job status, educational level, marital status, relationship to the PLWD, average hours of care per week, and living arrangements (whether they are staying with the PLWD under the same roof).
  Specific information about the care-recipients' characteristics and illness-related information of the PLWD will also be obtained: age, gender, existence of official diagnosis, type of dementia, and time since diagnosis.
Program Acceptability | 3 months
  A series of semi-structured interviews will be conducted with participants from the iSupport web-based intervention group, evaluating aspects such as: 1) motivation to participate; 2) user experience and barriers; 3) satisfaction with content, interface design and features; 4) program endorsement; and 5) any inconvenience / harm related to the study procedure (e.g. too many questionnaires, reasons for dropping out). Thematic analysis will be used to code the transcripts and derive themes.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Joey Loh, MPsych, Principal Investigator — Sunway University; Alvin Lai Oon Ng, DPsych, Principal Investigator — Sunway University
Locations (4):
- Malaysia (4):
  - University Malaya Medical Centre, Selangor, Petaling Jaya, Kuala Lumpur
  - Sarawak Heart Centre, Kota Samarahan, Sarawak
  - Sarawak General Hospital, Kuching, Sarawak
  - Sunway University, Subang Jaya, Selangor

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data that underlie the final results reported in the article (text, tables, figures, and appendices).
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Interested researchers should submit a reasonable request to the corresponding author (alvinn@sunway.edu.my). The requestor will need to sign a data access agreement that agrees to use the data solely for reasons outlined in the request.

REFERENCES:
- [Background] Loh KJ, Ng ALO, Chia YC, Lee WL, Mohan D, Renganathan E. Caring for people living with dementia and their informal caregivers: Current perspectives in Malaysia. Malays Fam Physician. 2024 Dec 27;19:69. doi: 10.51866/cm.674. eCollection 2024. PMID 39780913
- See also: World Health Organisation (2019). iSupport for Dementia: Training and support manual for carers of people with dementia. — https://www.who.int/publications/i/item/9789241515863